CLINICAL TRIAL: NCT02963727
Title: Knee Osteoarthrosis (KOA) in Jordanian Patients: a Phase I Dose-finding Study Using Wharton Jelly Derived Mesenchymal Stem Cells (WJMSC) for Advanced Stage III and IV KOA
Brief Title: Use of Wharton Jelly Derived Mesenchymal Stem Cells for Knee Osteoarthrosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanan Jafar (Other)
Responsible Party: Sponsor-Investigator, Hanan Jafar, Researcher, University of Jordan
Organization: University of Jordan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlloKneeUJCTC
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Knee Osteoarthrosis
Keywords: osteoarthrosis; Knee; Wharton Jelly
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wharton Jelly mesenchymal stem cell (Experimental): Intra-articular Wharton Jelly derived mesenchymal stem cell injection will be given for each patient in 2 doses, 50 million of WJMSC in each dose
  Interventions: Biological: Wharton Jelly derived mesenchymal stem cell

INTERVENTIONS:
Biological: Wharton Jelly derived mesenchymal stem cell — Intra-articular Wharton Jelly derived mesenchymal stem cell injection.

SUMMARY:
Wharton Jelly derived Mesenchymal Stem Cells (WJMSC) will be injected in patients diagnosed with Knee osteoarthrosis

DETAILED DESCRIPTION:
Ten patients from both genders diagnosed with Knee osteoarthrosis, will be enrolled according to strict inclusion and exclusion criteria. These patients will be injected with Wharton Jelly derived Mesenchymal Stem Cells. Then, they are followed by clinical assessment, laboratory investigations as well as magnetic resonance imaging (MRI) of the injected knee.

ELIGIBILITY:
Inclusion Criteria:

* Severe KOA stage III or IV by Laurance & Kellgren staging as judged by Posterioranterior (PA) Xray of the knee joint.
* Willing to participate by signing the informed consent

Exclusion Criteria:

1. Sublaxation beyond 20 degrees of the bones of the knee joint
2. Oral anticoagulants or heparin therapy
3. Heart failure or arrhythmia
4. Body Mass Index > 35
5. Uncontrolled Diabetes Mellitus.
6. Evidence of Infectious Diseases.
7. Active infection
8. Malignancy
9. Pregnancy
10. Anemia less than 11g/dl or thrombocytopenia less than 100,000 or leucopenia less than 3000.
11. Unreliable patients
12. Non-resident in Jordan

Ages: 42 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of the intra articular injection | 6 months
  patients will be monitored for any adverse events resulting from the intraarticular injection of WJMSC

SECONDARY OUTCOMES:
Assessment of the efficacy of intra-articular injection of WJMSC | 12 months
  The efficacy of the intra-articular injection of WJMSC will be assessed by Magnetic Resonance Imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided